CLINICAL TRIAL: NCT05875402
Title: Exploratory Clinical Trial on the Safety, Tolerability, Efficacy, and Pharmacokinetics of XKDCT080 in GCC-positive Recurrent or Refractory Solid Tumors With Single Center, Single Arm, and Dose Escalation
Brief Title: XKDCT080 in GCC-positive Recurrent or Refractory Solid Tumors With Single Center, Single Arm, and Dose Escalation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, wangjing, chief physician, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XKDCT080
Record Dates: First submitted 2023-04-25; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Colon Cancer
Keywords: Chimeric Antigen
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XKDCT080 treatment for patients with GCC target positivity (Experimental): Drug: XKDCT080 (chimeric antigen receptor T cell preparation targeting GCC)
  Dosage form: Cell suspension
  Dose: 30-50mL/bag
  Medication method: intravenous drip
  Frequency: Once
  Interventions: Drug: Chimeric antigen receptor T cell preparation targeting GCC

INTERVENTIONS:
Drug: Chimeric antigen receptor T cell preparation targeting GCC — Chimeric antigen receptor T cell preparation targeting GCC

SUMMARY:
The goal of this clinical trial is to assessing the safety and tolerability of XKDCT080 cells against recurrent or refractory solid tumors with GCC positivity.This experiment proposes to enroll 9-18 patients, the experimental drug is a chimeric antigen receptor T cell preparation targeting GCC.

Secondary purpose of the study

1. Evaluate the pharmacokinetic characteristics of XKDCT080 cells after intravenous infusion into GCC-positive patients with recurrent or refractory solid tumors;
2. Preliminary Evaluation of the Effectiveness of XKDCT080 Cells in Patients with Recurrent or Refractory Solid Tumors Positive for GCC;
3. Explore the relationship between cytokines and therapeutic efficacy in patients with recurrent or refractory solid tumors who are positive for GCC after intravenous infusion of XKDCT080 cells.

DETAILED DESCRIPTION:
This study adopts a single arm, single center, and dose increasing design, using a "3+3" design for dose increasing to evaluate the safety, tolerance, and effectiveness of XKDCT080 cells, as well as to evaluate the pharmacokinetic characteristics of XKDCT080 cells, the correlation between cytokines and efficacy, and immunogenicity.

The experimental process of this study is divided into seven stages: screening period, blood collection period, baseline period, clearance period, study treatment and safety observation period after treatment, follow-up period, and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients must meet ALL of the following criteria prior to participation:

  1. Age range from 18 to 75 years (including threshold), regardless of gender；
  2. Solid tumors with positive expression of guanylate cyclase (GCC) were detected by immunohistochemistry in tumor tissue；
  3. Patients with solid tumors who have failed standard treatment, are intolerant to standard treatment, have no standard treatment options, or have relapsed；
  4. At least one measurable lesion (non lymph node lesion with a length diameter of ≥ 10mm and lymph node lesion with a short diameter of ≥ 15mm) is required using the RECIST 1.1 standard；
  5. ECOG physical condition score 0-2；
  6. Blood routine standard: hemoglobin ≥ 90g/L (no blood transfusion within 14 days), neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 80 × 109/L；
  7. Blood biochemistry should meet the following standards: total bilirubin ≤ 1.5 × ULN (upper limit of normal value), ALT and AST ≤ 2.5 × ULN (excluding patients with liver metastasis); ALT and AST ≤ 5 in patients with liver metastasis × ULN； Serum creatinine ≤ 1 × ULN, glomerular filtration rate>50mL/min (GFR=[(140 age) × weight × (0.85 female)]/(72 × Scr), serum lipase and amylase<1.5 × ULN (upper limit of normal value), albumin ≥ 2.8g/dL;
  8. Cardiac ejection fraction>50%；
  9. No hemorrhagic diseases or coagulation disorders；
  10. The expected survival period is ≥ 12 weeks；
  11. The subjects voluntarily participated in the study and signed an informed consent form.

Exclusion Criteria:

* Patients with any of the following criteria will not be allowed to participation:

  1. Pregnant or lactating women;
  2. Participate in other drug clinical trials within 4 weeks before screening;
  3. There are uncontrollable cardiovascular and cerebrovascular diseases within the first 6 months of screening, such as heart failure or others;
  4. Have a history of drug abuse and are unable to quit or have a history of mental disorders;
  5. Has received any immune cell therapy in the past;
  6. Fungi, bacteria, viruses, or other infections that cannot be controlled or require antibiotic treatment;
  7. Hepatitis B surface antigen (HBsAg) positive or hepatitis B core antibody (HBcAb) positive, and HBV-DNA>500 IU/mL; Patients with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA; People who are positive for human immunodeficiency virus (HIV) antibodies; Syphilis antibody positive individuals;
  8. Allergies or intolerance to research drugs such as Tozumab, Fludarabine, Cyclophosphamide, Capecitabine, and other gonorrhea clearing drugs selected by the researchers;
  9. Active autoimmune diseases such as systemic lupus erythematosus or others within the first 3 months of screening;
  10. Suffering from known symptomatic central nervous system (CNS) diseases;
  11. The surgery was performed within 2 weeks before the single collection and the researcher believes that it may affect the safety of patient safety;
  12. There was a history of deep vein thrombosis or pulmonary embolism 6 months before enrollment;
  13. Used drugs that affect immune function one month before screening;
  14. Previously received GCC targeted therapy;
  15. According to the judgment of the researcher, patients who are not suitable to participate in this study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | 12 months]
  To characterize the safety profile of XKDCT080 in patients with advanced solid tumor as assessed by incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: jing wang, MD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No